CLINICAL TRIAL: NCT05842369
Title: Comparison of Two Approved Dialysis Methods for Treatment of Metabolic or Mixed Acidosis in Critically Ill Patients With Acute Kidney Injury and Indication for Renal Replacement Therapy
Brief Title: ADVOS® Versus CVVHD in Metabolic or Mixed Acidosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ADVOS-Acidosis UKE
Record Dates: First submitted 2023-04-02; First posted 2023-05-06 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Metabolic Acidosis
Keywords: acidosis; dialysis; acute kidney injury; renal replacement therapy; intensive care medicine; ADVOS
MeSH Terms: conditions — Acidosis; Acute Kidney Injury | interventions — Continuous Renal Replacement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ADVOS (Experimental): Application of the ADVOS device for
  Interventions: Device: ADVOS
- CVVHD (Active Comparator): Application of CVVHD
  Interventions: Device: CVVHD

INTERVENTIONS:
Device: ADVOS — Modulation of acid-base regulation in patients with acute kidney injury, meta- bolic or mixed acidosis and indication for renal replacement therapy
  Other Names: ADVOS® device; ADVITOS
  Arms: ADVOS
Device: CVVHD — Modulation of acid-base regulation in patients with acute kidney injury, meta- bolic or mixed acidosis and indication for renal replacement therapy
  Other Names: multiFiltrate / multiFiltratePRO
  Arms: CVVHD

SUMMARY:
The aim of the study is to investigate the effects of ADVOS® therapy in critically ill patients with acute kidney injury, necessity of renal replacement therapy and acidosis.

The investigators aim at assessing superiority of ADVOS® versus CVVHD for the primary outcome hours alive with normal pH (arterial pH ≤ 7,35) until 24 hours in a modified intention-to-treat analysis (mITT: replacement if dropped out before treatment start).

DETAILED DESCRIPTION:
Acute kidney injury (AKI) is frequently seen in patients treated at intensive care unit (ICU) and is associated with high morbidity and mortality. AKI occurs in more than 30% of critically ill patients. Various definitions for AKI have been used in the last decades, as a consequence reported incidence rates vary considerably from 13 to 78% in critically ill patients. AKI reflects a broad spectrum of clinical presentations, ranging from mild to se-vere injury, which may result in permanent loss of renal function. AKI is generally detected by a decrease in urine output (oliguria, anuria) and by an increase of renal serum markers (creatinine, blood-urea-nitrogen) with subsequent disorders in electrolyte homeostasis (e.g. hyperkalemia) and acid-base-regulation by means of metabolic acidosis. The AKIN criteria are well established criteria for diagnosis of AKI.

Different factors have been associated with development of AKI in critically ill patients. Age and pre-existing comorbidities are risk factors for development of AKI. Furthermore, infection and sepsis seem to be a mayor trigger for AKI. More than 50% of patients with septic shock develop AKI. Besides this radiocontrast agents, rapid progressive glomerulonephritis, rhabdomyolysis, trauma, circulatory shock, cardiac surgery, major non-cardiac surgery, nephrotoxic drugs and other causes are capable inducing AKI.

Metabolic acidosis, a frequent finding in AKI, is diagnosed when serum pH is reduced (pH < 7,35) and serum bicarbonate levels are abnormally low. Three major mechanisms lead to metabolic acidosis: 1) increased acid generation 2) loss of bicarbonate 3) decreased renal acid excretion. In AKI reduction of urine output and dimi-nished renal acid excretion results in subsequent metabolic acidosis.

Typical indications for renal replacement therapy (RRT) are hyperkalaemia, severe metabolic acidosis, diuretic-resistant volume overload, oliguria, anuria, uremic complications and some drug intoxications.

The use of RRT in Intensive Care Unit (ICU) patients increased over the last decades. In ICU setting continuous renal replacement therapies (CRRT) like continuous veno-venous hemodialysis (CVVHD) and continuous veno-venous hemodiafiltration are frequently used. Especially haemodynamic unstable patients benefit from CRRT compared to intermittent hemodialysis. Exact timing of starting CRRT and optimal intensity is still unk-nown.

The ADVOS device is a newly developed dialysis system based on the use of recycled albumin dialysate. The system has shown a high detoxification capacity in in-vitro and preclinical studies. The ADVOS procedure com-bines various therapeutic features that might be beneficial for patients with AKI. The ADVOS® device is capab-le to correct acid-base disorders like metabolic acidosis. Recent studies demonstrated a strong potential of correction of acidosis in critically ill patients suffering from multiorgan failure. Although the device is approved, there is a lack of clinical studies comparing of its effect on acidosis versus to other dialysis devices, that all can be used during clinical routine according to its indication.

ELIGIBILITY:
Inclusion Criteria:

* Metabolic or mixed acidosis with pH ≤ 7.25 and base excess ≤ -6 mmol/l
* Age ≥ 18 years
* Acute kidney injury with need for Renal Replacement Therapy (RRT)

Exclusion Criteria:

* Pregnancy
* Wards of the state/Prisoners
* Expected survival of less than 24 hours
* Contraindication for citrate anticoagulation
* Extracorporeal membrane oxygenation (ECMO)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2023-04-17 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Hours alive with normal pH (≥ 7.35) within first 24 hours of therapy | First 24 hours after initiation of study-specific therapy
  pH values are measured to determine acidaemia in critically ill patients. As defined by the study protocol, pH ≤ 7.25 and base excess ≤ -6 mmol/l are required to diagnose metabolic or mixed acidosis. Normalisation of pH (defined as ≥ 7.35, representing the lower margin of the pyhsiological pH range) is used as a surrogate marker for reversal of acedaemia and, thereby, device effectiveness. The time (hours) alive within the defined physiological range after initiation of therapy in the first 24 hours will be used to compare the intervention and control group.

SECONDARY OUTCOMES:
Time to first pH normalisation (≥ 7.35) | First 24 hours after initiation of study-specific therapy
  pH values are measured to determine azidemia in critically ill patients. As defined by the study protocol, pH ≤ 7.25 and base excess ≤ -6 mmol/l are required to diagnose metabolic or mixed acidosis. Normalisation of pH (defined as ≥ 7.35, representing the lower margin of the pyhsiological pH range) is used as a surragate marker for reversal of acedaemia and, thereby, device effectiveness. The time (hours) until reaching the defined physiological range for the first time will be used to compare the intervention and control group.
Days free of mechanical ventilation within the first 28d after randomization | From start of study-specific therapy until day 28
  Days free of mechanical ventilation across 28 days is used to compare the respiratory outcome between intervention and control group.
Days free of vasopressor therapy within the first 28d after randomization | From initiation of study-specific therapy until day 28
  Days free of vasopressor therapy within the first 28 days after randomization are used as surrogate marker to compare sepsis/vasoplegia reversal between intervention and control group.
Days free of renal replacement therapy within the first 28d after randomization | Assessment at baseline, days 1, 2, 3, 7, 14, 21, 28 as long as patient is still on intensive care unit
  Days free of renal replacement therapy within the first 28 days after randomization are used as an indicator of renal organ failure. Need for and length of renal replacement therapy is a prognostic factor in critically ill intensive care patients.
Course of severity of organ failure | Assessment at baseline, days 1, 2, 3, 7, 14, 21, 28 as long as patient is still on intensive care unit
  Severity of organ failures will be assessed on a daily basis using the Sequential Organ Failure Assessment (SOFA)-Score. Possible scores range from 0 to 24 points, whereby a higher score indicates a higher degree of organ failure.
Course of arterial blood gases | Time points Baseline, 0.5, 1, 2, 4, 6, 8, 12, 16, 20, 24, 48, 72 hours. If patient is still on intensive care unit, also on day 7, 14, 28
  The dynamics of arterial blood gases will be used to compare the intervention and control group.
Course of systemic hemodynamics | Timepoints Baseline, 0.5, 1, 2, 4, 6, 8, 12, 16, 20, 24, 48, 72 hours. If patient is still on intensive care unit, also on day 7, 14, 28
  The course of systemic haemodynamics is determined on the basis of vital parameters (e.g. mean arterial blood pressure, heart rate) as well as volume administration and catecholamine therapy will be used to compare the intervention and control group.
Intensive Care Unit and hospital length of stay | Assessment of status on day 28 and day 90
  Time point for discharge from intensive care unit and hospital stay
28 days and 90 days mortality | Assessment of status on day 28 and day 90
  Comparison of 28- as well as 90-day mortality between the study arms
Requirement and number of transfusions during ICU | Cumulative assessment until day 28 or end of intensive care unit stay, whichever comes first.
  The number of transfusions during ICU stay as well as the reason for need.
Biomarkers (i.e. markers of inflammation, coagulation, endothelial function, metabolism, drug monitoring) | Assessment at Baseline and time points 4, 16, 24, 48, 72 hours after initiation of study specific therapy as well as on day 7 and 28, if patient is still on intensive care unit
  Analysis of the changes in different biomarkers during the study-specific therapy to compare the two study groups up to day 28 or the transfer of metabolism, drug monitoring)

CONTACTS AND LOCATIONS:
Overall Officials: Olaf Boenisch, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- University Medical Center Hamburg-Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No